CLINICAL TRIAL: NCT04141280
Title: Study on the Material Basis of Syndromes of Insomnia and the Correlation Between
Brief Title: Study on the Material Basis of Syndromes of Insomnia and the Correlation Between Infrared Image
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Jun Song, director of science and education department, China Academy of Chinese Medical Sciences
Other Study IDs: ZZ2018015
Record Dates: First submitted 2019-10-19; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Insomnia
Keywords: Insomnia; Syndrome; Material basis; Infrared image; Relativity
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — the whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Insomnia group: According to the inclusion and exclusion criteria, 150 patients with insomnia were selected, which were divided into five groups: liver stagnation fire syndrome, phlegm heat syndrome, yin deficiency fire dysfunction syndrome, heart spleen deficiency syndrome and heart deficiency biliary syndrome.
- Normal group: According to the inclusion and exclusion criteria, 30 normal people were selected.

SUMMARY:
This study combined the insomnia syndrome with PSG, fMRI, neuroactive substance detection, and infrared heat map, observing the electrophysiological changes of insomnia patients with different syndromes,localizing brain function excitation zone and changes in neuroactive substances,and the response of the visceral function to the infrared Image，which reveal the biological material basis of insomnia syndrome, and analyze it's correlation with infrared Image, providing a scientific, objective and visual technical method for TCM diagnosis and treatment of insomnia.

DETAILED DESCRIPTION:
Insomnia belongs to the category of "Bu Mei" in Traditional Chinese Medicine(TCM). Long-term insomnia can increase the risk of heart disease, high blood pressure, senile dementia, anxiety, and depression. Therefore, the insomnia sparked a heated discussion in medical research.

It has a good effect in treating insomnia with TCM,but there are problems such as strong subjectivity of syndrome differentiation and large difference in efficacy between doctors.

The previous study found that the infrared Image reflects the visceral function of insomnia patients to a certain extent.Modern studies have shown that insomnia is closely related to the dysfunction of functional coordination between the brain's sleep and the arousal center, and neuroactive substances played an important role on it."Syndrome" is the key of clinical diagnosis and treatment of TCM. Investigators believe that the central nervous system imbalance of different syndrome of insomnia has a certain correlation with the infrared Image.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia group

  1. Meets the diagnostic criteria for ICSD-3 chronic insomnia;
  2. PSQI total score >16 points;
  3. Age 18-80 years old;
  4. Subjects agree with participate the research;
  5. Meets diagnostic criteria for five syndrome types of Chinese medicine insomnia.
* Normal group:

  1. Subjects had no insomnia or lacked of sleep in the past month.
  2. Blood pressure, blood sugar, and blood lipids are normal;
  3. Age 18-80 years old;
  4. Subjects agree with participate the research.

Exclusion Criteria:

* Insomnia group

  1. Suffering from serious neurological and psychiatric diseases;
  2. Suffering from systemic immune diseases, blood system diseases and obvious skin diseases;
  3. Having obvious symptoms of coronary heart disease and cerebrovascular disease;
  4. fMRI examination contraindications, including those who have undergone cardiac pacemaker implantation, those with grafts or metal foreign bodies, claustrophobia, etc.
  5. Unable to complete the tester.
* Normal group:

  1. PSQI total score ≥ 7 points；
  2. People who have taken drugs that affect sleep in the past week.
  3. Suffering from serious neurological and psychiatric diseases;
  4. Suffering from systemic immune diseases, blood system diseases and obvious skin diseases;
  5. Having obvious symptoms of coronary heart disease and cerebrovascular .
  6. fMRI examination contraindications, including those who have undergone cardiac pacemaker implantation, those with grafts or metal foreign bodies, claustrophobia, etc.
  7. Unable to complete the tester.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: After recruitment, subjects were collected from the clinic of China Academy of Chinese Medical Sciences and Xiyuan Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-10-20 (Estimated); Primary Completion 2021-10-20 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Four diagnostic information of Traditional Chinese Medicine(TCM) | 20 minutes
  All subjects filled in the form about the four diagnostic information of TCM in order to observe the subject's symptoms and judge the syndrome.
polysomnography | 9hours
  All subjects wore the polysomnography monitor electrodes and the data were record.According to physiological signal,observing the sleep structure and comparing the difference between the two groups.
fMRI | 30 minutes
  Detecting brain excitation functional area blood oxygen concentration and comparing the difference between the two groups.
Neuroactive substance detection | 9hours
  Blood is taken once before bedtime and the next morning in order to detect neuroactive substance,such as GABA,Glu,NE and so on.
Infrared image | 3 hours
  All subjects were completely exposed to the body in a closed room and tested infrared imaging technology.Observing the thermal state ΔT of each location or region of the subject, that is, the difference between the temperature of the trunk heat map and the mean temperature of the body surface.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index | 10minutes
  Pittsburgh sleep quality index（PSQI）is used to evaluate sleep quality of subjects.It's maximum is 21.The higher the score, the worse the sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Hongtao Lei, Study Director — Eperimental Research Center,China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel.Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Liu K, Kim J, Kim DW, Zhang YS, Bao H, Denaxa M, Lim SA, Kim E, Liu C, Wickersham IR, Pachnis V, Hattar S, Song J, Brown SP, Blackshaw S. Lhx6-positive GABA-releasing neurons of the zona incerta promote sleep. Nature. 2017 Aug 31;548(7669):582-587. doi: 10.1038/nature23663. Epub 2017 Aug 23. PMID 28847002
- [Background] Blackmer AB, Feinstein JA. Management of Sleep Disorders in Children With Neurodevelopmental Disorders: A Review. Pharmacotherapy. 2016 Jan;36(1):84-98. doi: 10.1002/phar.1686. PMID 26799351
- [Background] Manfridi A, Brambilla D, Mancia M. Sleep is differently modulated by basal forebrain GABA(A) and GABA(B) receptors. Am J Physiol Regul Integr Comp Physiol. 2001 Jul;281(1):R170-5. doi: 10.1152/ajpregu.2001.281.1.R170. PMID 11404291
- [Background] Basner M, Rao H, Goel N, Dinges DF. Sleep deprivation and neurobehavioral dynamics. Curr Opin Neurobiol. 2013 Oct;23(5):854-63. doi: 10.1016/j.conb.2013.02.008. Epub 2013 Mar 20. PMID 23523374